CLINICAL TRIAL: NCT01129180
Title: Phase I Dose-Escalation Study of Azacitidine (Vidaza) and Bortezomib (Velcade) in T-Cell Lymphoma
Brief Title: Bortezomib and Azacitidine in Treating Patients With Relapsed or Refractory T-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierluigi Porcu (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pierluigi Porcu, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08067; NCI-2010-01081 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2010-05-17; First posted 2010-05-24 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Peripheral T-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Prolymphocytic Leukemia; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Small Intestine Lymphoma; T-cell Large Granular Lymphocyte Leukemia
Keywords: T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral; Leukemia, Prolymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Large Granular Lymphocytic; Lymphoma, T-Cell | interventions — Azacitidine; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive bortezomib IV on days 4, 8, 11, and 15 and azacitidine SC on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity. Attempt to collect Correlative studies will be made.
  Interventions: Drug: azacitidine; Drug: bortezomib; Procedure: Correlative studies

INTERVENTIONS:
Drug: azacitidine — Given SC
  Other Names: 5-AC; 5-azacytidine; 5-AZC; azacytidine; ladakamycin; Vidaza
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Procedure: Correlative studies — Correlative studies will be collected pre-treatment, day 4 , day 15, day 29(pre-cycle 2)
  Other Names: PK; PD; pharmacodynamic; pharmacokinectic; laboratory biomarker analysis

SUMMARY:
RATIONALE: Bortezomib and azacitidine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with azacitidine in treating patients with relapsed or refractory T-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To determine the maximum tolerated dose (MTD) of VELCADE (BORTEZOMIB) in combination with Azacitidine in patients with relapsed/refractory CTCL/PTCL.

II. To define the specific toxicities and the dose-limiting toxicity (DLT) of VELCADE (BORTEZOMIB) in combination with Azacitidine.

SECONDARY OBJECTIVES I. To determine the overall response rate (ORR). II. To correlate the biological activity of Azacitidine as a demethylating agent (changes in target gene methylation and gene expression, DNMT1 protein expression, global methylation) with clinical endpoints and plasma pharmacokinetics of Azacitidine.

III. To characterize the biological activity of VELCADE (BORTEZOMIB) as a potential demethylating agent.

IV. To correlate intracellular concentration of Azacitidine-triphosphate with global DNA methylation and other biological endpoints as well as clinical response.

V. To explore the biologic role of microRNAs in determining clinical response to the VELCADE (BORTEZOMIB) plus Azacitidine combination and achievement of the other pharmacodynamic endpoints.

OUTLINE: This is a dose-escalation study of bortezomib.

Patients receive bortezomib IV on days 4, 8, 11, and 15 and azacitidine subcutaneously (SC) on days 1-5. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically documented T-cell lymphoma belonging to one of the following WHO entities: Peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS); Mycosis Fungoides and Sezary Syndrome (MF-SS); Angioimmunoblastic T-cell lymphoma (AITL); CD30-positive Anaplastic Large Cell Lymphoma (ALCL), systemic; T/NK-cell lymphoma, extranodal, nasal and nasal type; Hepatosplenic T-cell lymphoma, gamma/delta or alpha/beta; Enteropathy-associated T-cell lymphoma (EATL); Adult T-cell Leukemia/Lymphoma (ATLL); Subcutaneous panniculitis-like T-cell lymphoma (SCPTCL); Blastic T/NK-cell lymphoma/leukemia (CD4+CD56+ Hematodermic Tumor); T/NK-cell post-transplant lymphoproliferative disorders (PTLD); Large Granular Lymphocyte (LGL) Leukemia; T-cell Prolymphocytic Leukemia (T-PLL)
* Patients must have relapsed or refractory TCL
* Patients must have failed at least one prior systemic therapy
* Life expectancy must be greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have adequate organ function as defined below:
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* AST(aspartate aminotransferase) < 2.0 x ULN
* ALT(Alanine transaminase) < 2.0 x ULN
* Serum creatinine < 1.5 ULN
* New York Heart Association Congestive Heart Failure (NYHA CHF) Class II or better
* Platelet count >= 75,000/mm^3 (unless due to disease) within 14 days before enrollment
* Absolute neutrophil count of >= 1,500/mm^3 within 14 days before enrollment
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; if the patient does not agree, the patient is not eligible; women must agree to not get pregnant for the duration of the study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform the PI or the Study Nurse immediately
* Ability to understand and willingness to sign the written informed consent document before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients receiving any other investigational agents or patients who have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system (CNS) malignancy
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic composition to Azacitidine or VELCADE (BORTEZOMIB) that are not easily managed; patients with hypersensitivity to VELCADE (BORTEZOMIB), boron, or mannitol
* Patients must not have previously received Azacitidine or VELCADE (BORTEZOMIB) for any disease
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; as infection is a common feature of TCL, patients with active infection are permitted to enroll provided that the infection is under control; myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Pregnant women or women who are breastfeeding are excluded from this study; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* HIV-positive patients are ineligible; all patients will be screened for HIV
* Patients with pre-existing Grade 2 or higher neuropathy within 14 days before enrollment or other serious neurologic toxicity that would significantly increase risk of complications from VELCADE (BORTEZOMIB) therapy are excluded
* Patients with active, advanced malignant solid tumors are excluded
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD) of bortezomib in combination with azacitidine | up to 28 days
Specific toxicities and the dose limiting toxicity (DLT) of bortezomib in combination with azacitidine as assessed by NCI CTCAE (Common Toxicity Criteria for Adverse Effects) v4.0 | up to 2 years

SECONDARY OUTCOMES:
Overall response rate | up to 2 years
Correlation of the biological activity of Azacitidine as a demethylating agent with clinical endpoints and plasma pharmacokinetics | up to 2 years
Biological activity of bortezomib as a potential demethylating agent | up to 2 years
Correlation of intracellular concentration of azacitidine-triphosphate with global DNA methylation and other biological endpoints as well as clinical response | up to 2 years
Biologic role of microRNAs in determining clinical response to the bortezomib plus azacitidine combination and achievement of the other pharmacodynamic endpoints | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Porcu, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu